CLINICAL TRIAL: NCT03329820
Title: Quality of Life and Health Utility of Patients With Chronic Hepatitis B Infections
Brief Title: Quality of Life and Health Utility of Patients With CHB Infections
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Head and Clinical Professor, The University of Hong Kong
Other Study IDs: HKCTR-151
Record Dates: First submitted 2017-10-24; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Chronic Hepatitis B Infection
Keywords: Chronic hepatitis B infection; Health-related quality of life; Cost-effectiveness; Treatment; Chinese
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1 Uncomplicated CHB: Patients with chronic CHB infections but normal liver function and without cirrhosis or hepatocellular carcinoma
- 2 CHB with impaired liver function (LF) or CC w/o tx: CHB with impaired liver function or compensated cirrhosis, not on anti-viral treatment
- 3 CHB with impaired LF or CC with tx: CHB with impaired liver function or compensated cirrhosis, on anti-viral treatment.
- 4 Decompensated cirrhosis: Patients with CHB infection and cirrhosis complicated by one or more of the following: variceal bleeding, hepatic encephalopathy or ascites.
- 5 Hepatocellular carcinoma: Patients with confirmed diagnosis of hepatocellular carcinoma

SUMMARY:
The aim of the study is to assess the health-related quality of life (HRQOL) and preference-based health utilities of chronic hepatitis B (CHB) carriers in different stages of illness. It will also estimate the cost-effectiveness of anti-viral treatments resulting from the prevention of the progression of disease from uncomplicated CHB carriers to cirrhosis and hepatocellular carcinoma (HCC).

The following hypotheses will be tested:

1. Patients with chronic hepatitis B virus (HBV) have poorer health-related quality of life (HRQOL) than the general population;
2. Patients with more severe stages of chronic HB infections have lower health related quality of life and health utility values;
3. Anti-viral treatment can improve the HRQOL and health utility for patients with CHB infections;
4. The cost-effectiveness of different treatments for chronic HBV infections can be directly compared in terms of cost/QALY gained.

DETAILED DESCRIPTION:
Design, Setting & Subjects: A cross-sectional study and biomathematical modelling will be carried out. In the cross-sectional study, patients known to CHB carriers will be identified from the registries of the Ap Lei Chau, Aberdeen and Sai Yung Pun General Outpatient Clinics and Queen Mary Hospital. The biomathematical modelling will use a simulated cohort of patients aged 18 or above with CHB infections who may receive treatment in Hong Kong. Published data on the benefit of anti-viral treatments and the cross-sectional study data on preference-based health utility values of different stages of CHB infections will be used to estimate the cost-effectiveness of different treatment strategies using Markov modelling.

Interventions: Each subject in the cross-sectional study will be interviewed. Five strategies for management of CHB infections: 1) No treatment, 2) Interferon monotherapy, 3) lamivudine monotherapy, 4) adefovir and 5) combined treatment of lamivudine and adefovir, will be tested in the biomathematical modelling,.

Main Outcome Measures: Health-related quality of life measured by the SF-36, preference-based health utilities measured by the SF-6D. quality adjusted life years (QALYs) and cost of different treatment strategies for HBV infection.

Hypothesis: HRQOL and health utilities of patients with different illness stages, and the QALYs gained and cost-effectiveness of different therapeutic strategies will be established. The results will provide information on the health burden of CHB infections, and evidence on the cost-effectiveness of anti-viral treatments in preventing disease progression can be directly compared.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included in the study if they:

1. Are 18 years and above in age;
2. Are known to be HBsAg positive for more than six months;
3. Can be classified into one of the following sages of liver diseases:

(i) Uncomplicated CHB: Patients with chronic CHB infections but normal liver function and without cirrhosis or HCC.

(ii) CHB with impaired liver function or compensated cirrhosis, not on anti-viral treatment.

(iii) CHB with impaired liver function or compensated cirrhosis, on anti-viral treatment.

(iv) Decompensated cirrhosis: Patients with CHB infection and cirrhosis complicated by one or more of the following: variceal bleeding, hepatic encephalopathy or ascites.

(v) Hepatocellular Carcinoma: Patients with confirmed diagnosis of HCC

d. Have given written consent to take part in the study.

Exclusion Criteria:

Subjects will be excluded from the study if they have one of the following:

1. Unable to understand and communicate in Chinese Language;
2. Known cognitive impairment;
3. Diagnosed end-stage non-hepatitis B related chronic illness such as terminal cancer;
4. Patients currently abusing alcohol (>30 units/week) or illegal drugs;
5. Co-infection with HIV, hepatitis C virus (HCV) or hepatitis D virus (HDV);
6. Post-liver transplant;
7. Refuse to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese adults with chroni hepatits B infection.
Sampling Method: Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
SF-36 Health-related quality of life scores | Baseline
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.

SECONDARY OUTCOMES:
SF-6D Preference-based health utilities | Baseline
  The Short Form-6 Dimension (SF-6D) is a widely used preference-based generic HRQOL measure with a multiattribute classification system consisting of six dimensions: physical functioning, role functioning, social functioning, pain, mental health, and vitality. Each dimension is composed of three to five levels. The SF-6D values range from 0.315 to 1, with higher scores indicating better HRQOL anchoring on the 0 (dead) to 1 (full health) scale.
Quality adjusted life years | Baseline
  To calculate QALYs under different anti-viral treatments that prevent progressions to cirrhosis and HCC, the life expectancy of a person with or without cirrhosis or HCC will be estimated, starting with the age of 18.
Costs of different treatment strategies for HBV infection | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Two Regional Hospitals, Hong Kong, Hong Kong